CLINICAL TRIAL: NCT04233541
Title: Frailty Status and Increased Risk for Falls: The Role of Anticholinergic Burden
Brief Title: Frailty Status and Increased Risk for Falls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Ilkin Naharci, Assoc.Prof., Saglik Bilimleri Universitesi
Other Study IDs: 2016/1648-463
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Frailty; Fall; Anticholinergic Toxicity
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fallers: Participants who reported one or more falls within the 12 months preceding the study consist the group of ''fallers''.
  Interventions: Diagnostic Test: Fall assessment
- Non-fallers: Participants with no fall history consist the group of ''non-fallers''
  Interventions: Diagnostic Test: Fall assessment

INTERVENTIONS:
Diagnostic Test: Fall assessment — Through a comprehensive geriatric assessment carried out by our geriatrician led multidisciplinary team we gather information about fall recalls consistent with the definition of landing on the floor or ground.

SUMMARY:
We hypothesized that the use of anticholinergic medications may precipitate falls differently by frailty status in older adults. Community-dwelling older subjects admitted to the Geriatrics Outpatient Clinic prospectively enter into the study. Frailty status is defined according to the Physical Frailty Phenotype. The drugs are categorized according to the ACB scale

DETAILED DESCRIPTION:
Previous studies have found that the use of drugs with anticholinergic properties relate to increased prevalence of falls in older women and men. Frailty is associated with serious health outcomes including falls, hip fractures, and death. Frailty can be a relevant target to investigate its association with the risk of falls among the users of drugs with anticholinergic properties. A recent evidence suggests that the interaction between being frail and adverse outcomes in older adults receiving polypharmacy or centrally acting drugs is complex and not straightforward across all frailty phenotypes.

We classify the participants frail if they met at least three of five criteria, while those having one or two criteria were pre-frail, and others were non-frail. We determine the anticholinergic burden by using the Anticholinergic Cognitive Burden (ACB) Scale developed by Boustani et al.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults

Exclusion Criteria:

* a history of dementia,
* current delirium or psychotic symptoms,
* taking antipsychotic medications,
* being functionally dependent to others,
* difficulty in communicating with the interviewer,
* terminal illness,
* being bedridden or wheelchair bound (≥2 weeks),
* difficulty in standing or walking,
* incomplete data

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older subjects admitted to the Geriatrics Outpatient Clinic
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fall assessment | 1-2 hours
  We will assess the association between anticholinergic burden (ACB) and falls based on frailty status among older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Tasci, Prof., Principal Investigator — Gulhane Faculty of Medicine & Gulhane Training and Research Hospital
Locations (1):
- Gulhane Faculty of Medicine & Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No